CLINICAL TRIAL: NCT06922695
Title: Pill-in-Pocket Oral Anticoagulation Responding to Atrial Fibrillation Episodes Guided by Continuous Rhythm Monitoring and Automated Smartphone Alerts
Brief Title: Responding to AF: Pill-in-Pocket Anticoagulation Guided by Automated Monitoring and Alerts
Acronym: RESPOND-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Tim Betts MD MBChB FRCP, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17913; IRAS ID 329237 (Other: HRA (Health Research Authority - United Kingdom)); CPMS 56479 (Other: NIHR (National Institute for Health and Care Research - United Kingdom)); 24/WS/0126 (Other: West of Scotland Research Ethics Service (United Kingdom))
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation (Prevention of Stroke)
Keywords: Atrial Fibrillation; Pill-in-pocket anticoagulation; Anticoagulation; As-required anticoagulation; Intermittent anticoagulation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pill-in-pocket anticoagulation (Experimental): Participants will stop their oral anticoagulation after a 30-day period free of AF episodes. After this, they will only take their anticoagulation in response to an episode of AF detected by their implantable cardiac monitor. The participants will receive an automated smartphone alert instructing them to commence their anticoagulation as soon as AF is detected.
  Interventions: Other: Pill-in-pocket anticoagulation

INTERVENTIONS:
Other: Pill-in-pocket anticoagulation — Participants will stop their oral anticoagulation after a 30-day period free of AF episodes. After this, they will only take their anticoagulation in response to an episode of AF detected by their implantable cardiac monitor. The participants will receive an automated smartphone alert instructing them to commence their anticoagulation as soon as AF is detected.
  Other Names: As-required anticoagulation; Intermittent anticoagulation

SUMMARY:
Atrial Fibrillation (AF) is the most common sustained cardiac arrhythmia, affecting 1-2 million people in the UK. AF is characterised by uncoordinated electrical activation and ineffective contraction of the upper cardiac chambers. AF can occur in temporary episodes, as in paroxysmal AF, or can be sustained continuously beyond 7 days' duration, as in persistent AF.

The most significant potential complication of AF is stroke caused by a blood clot (thromboembolic stroke). If untreated, the risk of stroke in AF can be increased as much as five-fold, depending on the presence of other risk factors.

The mechanism of thromboembolic stroke in AF patients is complicated and understanding of factors involved remains incomplete. AF has been shown to disrupt normal bodily mechanisms for controlling bleeding and clotting (haemostasis) and normal blood flow inside the cardiac chambers. In disrupting these mechanisms, AF can be said to create a 'prothrombotic' state or environment within the blood and heart (a tendency to form clots) which can lead to blood clot formation and subsequently to stroke.

There is research evidence that AF-related stroke risk is not fixed and changes over time. This dynamic risk may be related to the episodic nature of AF, with stroke risk changing during an episode of AF and for a period of weeks after the episode terminates.

Analytic studies have shown that the risk of stroke is highest in the days after an AF episode has occurred, peaking at 5 days and returning to baseline by 30 days. Other studies have shown that the duration of the AF episode can also influence the risk of stroke following each episode, with longer episodes being higher risk.

This dynamic risk likely relates to changes in the activation of the body's blood-clotting system and changes in blood flow within the heart.

Current clinical guidelines recommend that patients with AF and risk factors for stroke are treated with daily, uninterrupted anticoagulation (blood-thinning medication) to reduce the risk of stroke. These guidelines do not take into account the temporal pattern of AF or the frequency or duration of AF episodes.

An emerging approach to anticoagulation in AF is pill-in-pocket oral anticoagulation (PIPOAC). In this approach, AF patients only take their anticoagulation in response to episodes of AF, and for a period of time after normal heart rhythm is restored. This approach may suit AF patients who have lower risk, lower frequency AF and who wish to reduce their exposure to anticoagulation medication. It may also suit AF patients who have higher bleeding risk related to anticoagulation.

The RESPOND-AF study proposes a novel approach to delivering PIPOAC. It is a pilot study of this novel approach recruiting 50 participants. This includes participants having continuous heart rhythm monitoring using the Medtronic LINQ II implantable cardiac monitor. The LINQ II continuously monitors for evidence of AF. If AF is detected a transmission is uploaded to the Medtronic Carelink cloud portal.

Traditionally, healthcare professionals need to sign in to this portal to check for any transmissions. For the purposes of PIPOAC this traditional approach would be too slow and create a burdensome workload for clinicians. Due to the properties of blood clot formation in AF, it is important to initiate oral anticoagulation within 48 hours of AF episode onset to disrupt the clot-formation process.

For the purposes of this study, the investigators have developed a custom-designed software which continuously screens for transmissions of AF on the Carelink cloud portal. When an AF episode has been detected by the LINQ II monitor, the software will send an SMS smartphone alert to the patient informing them of the AF episode and instructing them to commence their oral anticoagulation as soon as possible. This approach, if shown to be safe and effective and acceptable to patients, could open the path to wider use of Pill-in-pocket oral anticoagulation.

This novel treatment can reduce the need for anticoagulation, meaning fewer bleeding complications. Pill-in-pocket oral anticoagulation empowers patients by offering a new treatment choice beyond current limited options.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the trial.
2. Understand the risk and willing to discontinue oral anticoagulation (OAC).
3. Any gender aged 18 years or above.
4. Non-valvular paroxysmal atrial or persistent atrial fibrillation (AF) with a current rhythm control strategy. Paroxysmal patients must have < 3 documented or symptomatic episodes of >1 hour duration in the previous 3 months. Persistent patients must have been in continuous sinus rhythm for at least 4 weeks prior to enrolment.
5. CHA2DS2-VASc score between 1 and 3 in men and between 2 and 4 in women.
6. Able to take direct-acting oral anticoagulant (DOAC) in guideline recommended doses.
7. Left atrial (LA) diameter on echocardiogram less than 5 cm (anteroposterior dimensions) or LA volume less than 48 ml/m2.

Exclusion Criteria:

1. Any contraindication to OAC therapy with a DOAC in guideline recommended doses.
2. Mechanical heart valve prosthesis or moderate-to-severe mitral valve stenosis.
3. Permanent atrial fibrillation.
4. Hypertrophic cardiomyopathy.
5. Documented previous thromboembolic event (stroke, transient ischaemic attack or systemic embolism).
6. Spontaneous echo contrast observed in any imaging modality.
7. History of intracardiac thrombi.
8. History of congenital heart disease.
9. Severe chronic renal disease (eGFR <15 ml/m) or on renal replacement therapy.
10. Pregnant or planning pregnancy.
11. Indication for OAC other than atrial fibrillation.
12. Inability to comply with protocol.
13. Smartphone with operating system (OS) not compatible with MyCareLink Heart app.
14. Contraindication for implantable cardiac monitor.
15. Visual or physical impairment that prevents ability to read and acknowledge smartphone/watch notifications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
To investigate the reduction in oral anticoagulation (OAC) utilisation during follow-up. | During follow-up (minimum 13 months)
  Calculate the proportion of time off anticoagulation OAC

SECONDARY OUTCOMES:
Thromboembolic events (Ischaemic stroke, transient ischaemic attack (TIA) and systemic embolism) | During follow-up (minimum 13 months)
  Calculate the rate of ischaemic stroke, TIA and systemic embolism in patients on as-required OAC
Major bleeding | During follow-up (minimum 13 months)
  Calculate the rate of major bleeding in patients on as-required OAC
Minor bleeding | During follow-up (minimum 13 months)
  Calculate the rate of minor bleeding in patients on as-required OAC
Any stroke (ischaemic, haemorrhagic or undetermined) | During follow-up (minimum 13 months)
  Calculate the stroke rate (ischaemic, haemorrhagic or undetermined)
All-cause mortality | During follow-up (minimum 13 months)
  Calculate the rate of all-cause mortality in patients on as-required OAC
Protocol adherence | During follow-up (minimum 13 months)
  Calculate the number of daily transmissions and percentage of patients that restarts OAC within 24 hours of the smartphone-alert.
To assess response time from AF episode onset to patient starting as-required OAC | During follow-up (minimum 13 months)
  Time from AF episode onset to detection, time to alerts being sent and acknowledged and OAC

CONTACTS AND LOCATIONS:
Overall Officials: Prof Tim R. Betts MD MBChB FRCP, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Trust, John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not included in Informed Consent Form.

DOCUMENTS (1):
  • Study Protocol (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT06922695/Prot_000.pdf